CLINICAL TRIAL: NCT05574413
Title: Impact of Acute Exercise Intensity and Pattern on Cytokine Function
Acronym: AEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AEX2022
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Inflammation
Keywords: Exercise; Cytokines; Leukocytes; Interleukin-10; Interleukin-6
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Repeated measures randomized counterbalanced crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resting (no exercise) control (Placebo Comparator): Resting (no exercise) control condition
  Interventions: Other: Resting (no exercise) control
- Moderate intensity continuous exercise (MICE) (Experimental): Experimental session involving an acute bout of moderate intensity continuous exercise (MICE; continous cycling expending 350 kcal at 70% of lactate threshold)
  Interventions: Other: Moderate intensity continuous exercise
- High intensity continuous exercise (HICE) (Experimental): Experimental session involving an acute bout of high intensity continuous exercise (HICE; continuous cycling expending 350 kcal at 10% of the difference between lactate threshold and VO2peak)
  Interventions: Other: High intensity continuous exercise
- High intensity interval exercise (HIIT) (Experimental): Experimental session involving an acute bout of high intensity interval exercise (HIIT; cycling intervals expending 350 kcal at 10% of the difference between lactate threshold and VO2peak)
  Interventions: Other: High intensity interval exercise

INTERVENTIONS:
Other: Moderate intensity continuous exercise — Participants will perform an acute bout of continuous cycling at 70% of the power output at lactate threshold until an energy expenditure of 350 kcal is achieved. Blood samples will be obtained immediately before and immediately, 30, and 90 minutes after exercise.
  Other Names: MICE
  Arms: Moderate intensity continuous exercise (MICE)
Other: High intensity continuous exercise — Participants will perform an acute bout of continuous cycling at 10% of the difference between lactate threshold and VO2peak until an energy expenditure of 350 kcal is achieved. Blood samples will be obtained immediately before and immediately, 30, and 90 minutes after exercise.
  Other Names: HICE
  Arms: High intensity continuous exercise (HICE)
Other: High intensity interval exercise — Participants will perform an acute bout of interval cycling at at 10% of the difference between lactate threshold and VO2peak until an energy expenditure of 350 kcal is achieved. Blood samples will be obtained immediately before and immediately, 30, and 90 minutes after exercise.
  Other Names: HIIE
  Arms: High intensity interval exercise (HIIT)
Other: Resting (no exercise) control — Participants will remain in a rested state (i.e., no exercise) for the entire session. Blood samples will be obtained at the same time-points as the exercise sessions.
  Other Names: CTL
  Arms: Resting (no exercise) control

SUMMARY:
The immune system helps prevent illness, fights off infections, and repairs damaged tissues following an injury. However, when immune cells remain active for prolonged periods of time - a state known as "chronic inflammation" - they can contribute to the development and progression of chronic diseases like heart disease and diabetes. Exercise can reduce the risk of developing many of these diseases and at least part of the health benefits of exercise are due to the ability of exercise to reduce "chronic inflammation". The inflammation-lowering effects of exercise are typically captured by measuring hormone-like molecules released from immune cells called "cytokines" in the blood. In addition to changes in circulating cytokine levels, exercise may also alter how immune cells respond to these cytokines. How exercise intensity (i.e., how hard you are working during exercise) and pattern (i.e., exercising as a long continuous bout or in short intervals) impact the ability of immune cells to respond to cytokines is not well understood. A better understanding of how exercise intensity and pattern of exercise for reducing chronic inflammation may help determine the best types of exercises for improving health and preventing chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age
* Body mass index between 18.5-30 kg/m^2
* Free of cardiometabolic and autoimmune/inflammatory disease

Exclusion Criteria:

* Competitive endurance athlete
* Cigarette smoker
* Currently taking immunomodulatory/anti-inflammatory medications
* Currently pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
IL-10 mediated STAT3 phosphorylation | Change from pre-exercise to immediately and 90-min post-exercise
  Ex vivo leukocyte STAT3 phosphorylation in response to IL-10 treatment

SECONDARY OUTCOMES:
IL-10 mediated TNF-alpha inhibition | Change from pre-exercise to immediately and 90-min post-exercise
  Ex vivo inhibition of TNF-alpha production in response to IL-10 treatment
IL-6 mediated STAT3 phosphorylation | Change from pre-exercise to immediately and 90-min post-exercise
  Ex vivo leukocyte STAT3 phosphorylation in response to IL-6 treatment
IL-6 mediated TNF-alpha inhibition | Change from pre-exercise to immediately and 90-min post-exercise
  Ex vivo inhibition of TNF-alpha production in response to IL-6 treatment
Plasma IL-10 | Change from pre-exercise to immediately, 30-, and 90-min post-exercise
  Concentration of IL-10 in plasma samples
Plasma IL-6 | Change from pre-exercise to immediately, 30-, and 90-min post-exercise
  Concentration of IL-6 in plasma samples
Plasma TNF-alpha | Change from pre-exercise to immediately, 30-, and 90-min post-exercise
  Concentration of TNF-alpha in plasma samples
Hematology panel | Change from pre-exercise to immediately, 30-, and 90-min post-exercise
  Complete blood count
Extracellular vesicles | Change from pre-exercise to immediately, 30-, and 90-min post-exercise
  Concentration of extracellular vesicles in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan P Little, PhD, Principal Investigator — UBC Okanagan
Locations (1):
- UBC Okanagan, Kelowna, British Columbia, Canada